CLINICAL TRIAL: NCT03898414
Title: Patterns and Outcome of Autoimmune Related Chronic Liver Disease : Retrospective Study
Brief Title: Patterns and Outcome of Autoimmune Related Liver Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yomna Hammam Abou El-Wafa, Resident, Assiut University
Other Study IDs: autoimmune liver disease
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Autoimmune Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the different patterns of autoimmune related chronic liver disease to assess the prevalence of various types and outcome of treatment of autoimmune related chronic liver disease

DETAILED DESCRIPTION:
Autoimmune liver diseases (AILD) are a group of immunologically induced hepatic damage that are either hepatocellular or cholestatic. The hepatocellular forms are characterized by a significant elevation of the serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST), as compared with the biliary enzymes,together with elevated serum bilirubin Autoimmune hepatitis (AIH) is the typical example of hepatocellular autoimmune liver diseases, but it can also be presented under a cholestatic pattern. Autoimmune hepatitis has a scoring diagnostic system and respond in most cases to the treatment with prednisolone and azathioprine. Primary biliary cirrhosis (PBC) is the second most common autoimmune liver diseases , with a cholestatic presentation and characterized by positive antimitochondrial antibody (AMA). It has an excellent response and long term outcome with the administration of ursodeoxycholic acid (UDCA) Another autoimmune liver disease that is thought to be a variant of PBC is the autoimmune cholangitis, being a disease that has biochemical and histological features similar to PBC; but the AMA is negative. Primary sclerosing cholangitis (PSC) is a rare entity of autoimmune liver disease that has a cholestatic presentation and respond poorly to the treatment, with the ultimate progression to advance liver cirrhosis in most patients Other forms of autoimmune liver disease include the overlap syndromes (OS), which are diseases with mixed immunological and histological patterns of two autoimmune liver disease the most commonly recognized one is AIH-PBC overlap (AIH-PSC overlap is less common). The treatment of OS involves the trial of ursodeoxycholic acid and different immunosuppressant.

The vast majority of studies examining the incidence and prevalence of autoimmune liver disease have focused on PBC. Estimates of both disease incidence and prevalence vary quite widely between studies of specific defined populations.

Primary biliary cirrhosis (PBC), autoimmune hepatitis (AIH) and primary sclerosing cholangitis (PSC) are chronic liver diseases that likely have an autoimmune basis to their pathogenesis. Although significant strides have been made in the clinical management of these conditions, their pathogenesis remains obscure. Understanding of various epidemiological factors may shed light on predisposing or causative factors of these diseases There are limited Egyptian studies available on prevalence and spectrum of autoimmune liver diseases in cholestatic liver diseases, so the investigators will design this work to evaluate the prevalence of autoimmune liver diseases in cholestatic liver diseases and clinical profile of the various autoimmune liver diseases.

ELIGIBILITY:
-Inclusion criteria :

Patients that will fulfill the following criteria will be enrolled:

1. Patients diagnosed as AIH According to the simplified criteria of AIH scoring
2. Patients diagnosed as PBC or PSC according to the Amiracan association of study of liver disease (AASLD) - For all enrolled patients the presentation, treatment history, and outcome of treatment will be evaluated.

Exclusion criteria :

1-- All patients with chronic liver disease other than autoimmune liver disease will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients 18-60 years old with autoimmune related chronic liver disease
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of patterns of autoimmune chronic liver diseases | 2013-2019
  Evaluation of patterns of autoimmune chronic liver diseasesupport and outcome of treagent of these diseases

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Abou Elwafa, Principal Investigator — Assiut University; Adnan Mohamed, Lecturer, Study Director — Assiut University; Mohamed Mekky, Ass. Prof., Study Director — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

REFERENCES:
- [Background] Lee YM, Teo EK, Ng TM, Khor C, Fock KM. Autoimmune hepatitis in Singapore: a rare syndrome affecting middle-aged women. J Gastroenterol Hepatol. 2001 Dec;16(12):1384-9. doi: 10.1046/j.1440-1746.2001.02646.x. PMID 11851837
- [Background] Floreani A, Niro G, Rosa Rizzotto E, Antoniazzi S, Ferrara F, Carderi I, Baldo V, Premoli A, Olivero F, Morello E, Durazzo M. Type I autoimmune hepatitis: clinical course and outcome in an Italian multicentre study. Aliment Pharmacol Ther. 2006 Oct 1;24(7):1051-7. doi: 10.1111/j.1365-2036.2006.03104.x. PMID 16984499
- [Background] Kumagi T, Alswat K, Hirschfield GM, Heathcote J. New insights into autoimmune liver diseases. Hepatol Res. 2008 Aug;38(8):745-61. doi: 10.1111/j.1872-034X.2008.00366.x. Epub 2008 May 7. PMID 18462376
- [Background] Fallatah HI, Akbar HO, Qari YA. Autoimmune hepatitis: Single-center experience of clinical presentation, response to treatment and prognosis in Saudi Arabia. Saudi J Gastroenterol. 2010 Apr-Jun;16(2):95-9. doi: 10.4103/1319-3767.61235. PMID 20339178
- [Background] Hirschfield GM, Al-Harthi N, Heathcote EJ. Current status of therapy in autoimmune liver disease. Therap Adv Gastroenterol. 2009 Jan;2(1):11-28. doi: 10.1177/1756283X08098966. PMID 21180531
- [Background] Bogdanos DP, Gershwin ME. What is new in primary biliary cirrhosis? Dig Dis. 2012;30 Suppl 1:20-31. doi: 10.1159/000341118. Epub 2012 Oct 11. PMID 23075865